CLINICAL TRIAL: NCT00599079
Title: Open, Noncomparative Trial of Azithromycin in the Treatment of M.Avium Complex (MAC) Lung Disease
Brief Title: Azithromycin in the Treatment of M. Avium Complex Lung Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at Tyler (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Richard J. Wallace, Jr., M.D., Chairman Department of Microbiology, The University of Texas Health Science Center at Tyler
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 340
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Mycobacterium Avium Complex Lung Disease
Keywords: MAC
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azithromycin (Experimental): Azithromycin combined with 2 other drugs given 3 times weekly for MAc lung disease
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Azithromycin Daily Dosage dependent on clinical factos such as age, weight and patient specific health descriptors
  Other Names: Zithromax

SUMMARY:
To determine the safety and efficacy of azithromycin in the treatment of lung infection with M.avium complex and M. abscessus lung disease.

DETAILED DESCRIPTION:
To study the safety and efficacy of azithromycin in combination treatment for M. abscessus and MAC lung disease

ELIGIBILITY:
Inclusion Criteria:

* Meet American Thoracic Society criteria for nontuberculous lung disease: two or more AFB smear positive, culture positive sputums or bronchoscopic samples and/or two or more AFB smear negative respiratory samples with moderate to heavy growth (2+-4+); abnormal CXR consistent with M. avium lung disease; abnormal CXR consistent with M. avium lung disease; absence of other lung pathogens (except for the coexistence of M. abscessus).
* Age 18 and older
* Pretreatment isolate of M. avium complex available for MIC determination

Exclusion Criteria:

* History of macrolide allergy
* Received macrolide therapy in last two months
* Children less than 18 years of age
* If a menstruating female, not pregnant and on adequate birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 1993-02 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Clinical and microbiological outcomes such as clinical symptoms and laboratory cultures | 6 months
  neg cultures X3( sputum conversion)

SECONDARY OUTCOMES:
Microbiological cultures | 1yr
  culture neg 1 yr on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Wallace Jr., M.D., Principal Investigator — The University of Texas Health Science Center at Tyler
Locations (1):
- The University of Texas Health Science Center at Tyler, Tyler, Texas, United States

IPD SHARING:
Plan to Share IPD: No